CLINICAL TRIAL: NCT02890524
Title: Effects of a Night Guard on Aphthous Stomatitis
Brief Title: Tokushima Night Guard for Recurrent Aphthous Stomatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tokushima (Other)
Responsible Party: Principal Investigator, Yasusei Kudo, Associate Professor, University of Tokushima
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Tokushima #2053
Record Dates: First submitted 2016-08-21; First posted 2016-09-07 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Aphthous Stomatitis
Keywords: aphthous stomatitis; night guard; inflammatory cytokine
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Night guard (Experimental): the night guard made of EVA
  Interventions: Device: night guard
- Placebo night guard (Placebo Comparator): Placebo night guard made of EVA
  Interventions: Device: placebo night guard

INTERVENTIONS:
Device: night guard — 60 days before and after intervention with the night guard
  Arms: Night guard
Device: placebo night guard — 60 days before and after intervention with the placebo night guard
  Arms: Placebo night guard

SUMMARY:
The investigators will investigate whether the night guard can suppress the development of recurrent aphthous stomatitis (RAS). The investigators will record the patients' oral condition for 60 days before and after intervention with the night guard made of Ethylene-Vinyl Acetate copolymer (EVA). The patients' saliva will be analyzed for measurement of inflammatory cytokines or oxidative stress.

DETAILED DESCRIPTION:
The study involved 20 patients (8 male and 12 female) with RAS. These patients suffered from RAS at least once a month. The investigators will record their oral condition for 60 days before and after intervention with the night guard made of EVA. Their saliva will be analyzed for further studies including measurement of inflammatory cytokines or oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered from recurrent aphthous stomatitis at least once a month

Exclusion Criteria:

* People do not have a experience of recurrent aphthous stomatitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
number of developed aphthous stomatitis | through study completion, an average of 1 year

SECONDARY OUTCOMES:
days until healing | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yasusei Kudo, DDS, PhD, Principal Investigator — Tokushima University
Locations (2):
- Japan (2):
  - Tada Dental Clinic, Kakogawa, Hyōgo
  - Tokushima University Hospital, Tokushima

IPD SHARING:
Plan to Share IPD: Undecided